CLINICAL TRIAL: NCT04930159
Title: Social Interventions for Support During Treatment for Endometrial Cancer and Recurrence
Acronym: SISTER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kemi Doll, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00012990; RG1121627 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2021-12773 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced usual care (No Intervention): Written materials in an appealing package.
- Facilitated group support (Active Comparator): Weekly group gatherings.
  Interventions: Behavioral: Facilitated group support
- 1:1 Peer Support (Active Comparator): Individual peer support calls.
  Interventions: Behavioral: 1:1 Peer Support

INTERVENTIONS:
Behavioral: Facilitated group support — Weekly group gatherings where content will alternate between group conversation and focused topics (e.g., treatment side-effects, mental health, family dynamics, nutrition, financial hardship) with facilitated discussion by a trained professional in nutrition, psychotherapy, cognitive behavioral therapy, or medicine. Each group will cycle through the same order of topics.
  Arms: Facilitated group support
Behavioral: 1:1 Peer Support — 1:1 peer support via telephone or video either during or near a treatment visit. Call content will be focused on social support and driven by the needs of the participant.
  Arms: 1:1 Peer Support

SUMMARY:
The SISTER study is a randomized trial, looking at various modalities of social support for Black patients undergoing treatment for endometrial cancer. There are three study arms: group support, 1:1 peer support, and enhanced usual care. The primary outcome is treatment completion, and the secondary outcome is social isolation.

DETAILED DESCRIPTION:
SISTER is a prospective, open randomized controlled trial of U.S. Black/African-American people with high-risk endometrial cancer requiring treatment with chemotherapy, radiation, or immunotherapy. We will compare social support interventions of enhanced usual care, weekly group-based support, and 1:1 peer support to determine the most effective option to improve treatment completion and decrease social isolation.

The SISTER study comparators are based on multiple systematic reviews of peer support literature, input from the multi-stakeholder Steering Group of the Endometrial Cancer Action Network for African Americans (ECANA), two focus groups of Black women with EC, and cancer center leadership at selected enrollment sites. The core function of each comparator is to decrease social isolation for women on active treatment. Of the peer support intervention options available, the SISTER study includes the two that have the most data collected among Black women with cancer, have been most efficacious with regard to social isolation9 and treatment completion, and were enthusiastically supported by ECANA patient partners and focus group data.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 years of age or older; and
2. Self-identify as Black/African American
3. Presenting with high-risk EC established by anatomic pathology as tumor stage and grade classification by the following:

   1. Pathology documentation from any hospital/clinic/medical center, and
   2. FIGO Stage 1A with Grade 2, Grade 3, or Grade 4 of any histology type or
   3. FIGO Stage 1A with non-endometrioid (carcinosarcoma, serous, clear cell, undifferentiated or mixed) histology
   4. FIGO Stage 1B, 2, 3, or 4 of any grade or histology
   5. Recurrent endometrial cancer of any stage or grade
4. Documented provider recommendation and patient plan to initiate adjuvant therapy with chemotherapy, radiation, and/or immunotherapy.

Exclusion Criteria:

Participants must not have any of the following exclusion criteria:

1. Newly diagnosis of FIGO Stage IA Grade 1 endometrioid adenocarcinoma
2. Previous history of other cancer diagnosis requiring chemotherapy, radiation therapy, or immunotherapy within the past 12 months;
3. Incarcerated in a detention facility or in police custody (patients wearing a monitoring device can be enrolled) at baseline/screening;
4. Contraindication to all non-surgical therapy available for endometrial cancer (i.e., chemotherapy, radiation, and immunotherapy contraindicated);
5. Enrollment into hospice prior to randomization
6. Unable to provide written informed consent in English;
7. Unable to be contacted for research surveys;
8. Recent hospitalization for psychiatric illness in the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Treatment completion (relative dose) | 6 months
  Relative dose is the ratio of actual-to-expected total dose of treatment received. The calculation of expected total dose will be made from the baseline treatment recommendation data collected at enrollment.

SECONDARY OUTCOMES:
Patient-reported social isolation (SPS-24) | 6 months
  The Social Provisions Scale (SPS) is one of the most frequently used scales on social support, and is validated to measure the components of social support that directly impact health outcomes: attachment, social integration, reassurance of worth, reliable alliance, guidance, and opportunity for nurturance.

CONTACTS AND LOCATIONS:
Overall Officials: Kemi M Doll, MD, MS, Principal Investigator — University of Washington
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Miami, Miami, Florida
  - The University of Chicago, Chicago, Illinois
  - Louisiana State University - New Orleans, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - MedStar Health Research Institute, Columbia, Maryland
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared with other researchers. Researchers will be required to receive approval from the SISTER Advocate Advisory Board to receive data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The time frame is to be determined, in partnership with the SISTER Executive Committee and Advocate Advisory Board
Access Criteria: The access criteria is to be determined, in partnership with the SISTER Executive Committee and Advocate Advisory Board

REFERENCES:
- [Derived] Oluloro A, Comstock B, Monsell SE, Gross M, Wolff EM, Sage L, Alson J, Lavallee DC, Hempstead B, Moore A, Katz R, Doll KM. Study Protocol for the Social Interventions for Support During Treatment for Endometrial Cancer and Recurrence (SISTER) study: a community engaged national randomized trial. J Comp Eff Res. 2024 Mar;13(3):e230159. doi: 10.57264/cer-2023-0159. Epub 2024 Feb 13. PMID 38348827